## A clinical prospective study to validate a risk scoring model for the hepatic metastases from gastric cancer after curative surgery (DJY003 Trail)

**Edition Number: 1.0** 

Edition Generation Date: Apr 29, 2023 Principal Investigator: Jingyu Deng

Research Institute: Cancer Hospital & Institute of Tianjin Medical University

ClinicalTrials.gov ID: NCT06023966

## **Protocol:**

- Curative gastrectomy and D2 lymphadenectomy
- Postoperative pathology confirmed gastric cancer without distant metastasis, distant lymph node metastasis or peritoneal dissemination (M0)
- Age between 18 and 70 years
- KPS score >60
- No liver occupying disease and other chronic diseases of the liver prior to curative surgery
- No seriously chronic diseases of important organs

